CLINICAL TRIAL: NCT00801905
Title: Effect of Topical Nepafenac in Macular Thickening Related to Pan-retinal Photocoagulation
Acronym: NEPAF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NEPAFENAC IN PRFC; NEPAFENACO
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Macular Thickening; Macular Edema
Keywords: Macular thickening; Macular edema; Pan-retinal photocoagulation; Nepafenac; Topical non-steroidal anti inflammatory agents
MeSH Terms: conditions — Macular Edema | interventions — nepafenac; Lubricants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Nepafenac (Active Comparator): Topical nepafenac 0.1% is administrated every 6 hour 1 week before start pan-retinal photocoagulation and 4 weeks during all laser session performed biweekly, and 4 weeks after last laser sessión was completed.
  Interventions: Drug: Nepafenac
- 2: placebo (Placebo Comparator): Topical lubricating is administrated every 6 hours at fellow eye 1 week before start pan-retinal photocoagulation, 4 weeks during each laser session performed biweekly, and 4 weeks after last laser sessión was completed
  Interventions: Other: Lubricant

INTERVENTIONS:
Drug: Nepafenac — Topical nepafenac 0.1% is administrated every 6 hour 1 week before start pan-retinal photocoagulation and 4 weeks during all laser session performed biweekly, and 4 weeks after last laser sessión was completed.
  Other Names: Nevanac 0.1%
  Arms: 1: Nepafenac
Other: Lubricant — Topical lubricating is administrated every 6 hours at fellow eye 1 week before start pan-retinal photocoagulation, 4 weeks during each laser session performed biweekly, and 4 weeks after last laser sessión was completed
  Other Names: Systane
  Arms: 2: placebo

SUMMARY:
The purpose of this study is to determine whether topical nepafenac (qid) is effective in preventing and treating macular thickening related pan-retinal photocoagulation in patients with diabetic retinopathy.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of topical nepafenac 0.1 %, in preventing and in treating macular thickening related to pan-retinal photocoagulation in diabetic patients. Material and methods: This is a prospective, longitudinal, and controlled study in patients with diabetic retinopathy (severe non-proliferative and proliferative retinopathy), with a symmetric severity in both eyes and without a clinical significant macular edema. The best corrected visual acuity (BCVA) in all patients was 20/80 or better. All patients will undergo pan-retinal photocoagulation in three different sessions (with 2 weeks in apart between them). Each patient will receive topical nepafenac 0.1% (qid) on one eye, and placebo (qid) at the fellow eye, starting 1 week before the first retinal photocoagulation session and continued for 9 weeks ( ending 4 weeks after pan-retinal photocoagulation is completed). Spectral domain OCT and BCVA in ETDRS scale will be performed before and at 2 weeks after each laser session, and at 1, 2 and 3 months after treatment completed. BCVA and OCT outcomes of each studied period will be compared on both eyes, and side effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Severe and proliferative Diabetic Retinopathy
* Symmetric severity grade on both eyes
* Best corrected visual acuity better than 20/80

Exclusion Criteria:

* Clinical significant macular edema
* Lens opacity
* Ocular surgery 6 months or less before recruit
* Uveitis history
* Actual use of topical or systemic non-steroidal anti inflammatory agents
* Actual or history of other macular diseases
* Ocular surface diseases
* Vitreomacular traction syndrome
* Other vascular retinal diseases different to diabetic retinopathy
* Actual or history of use of topical prostaglandin analogues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Central macular thickening | 2 weeks after each laser session and 1 and 2 months after last laser session

SECONDARY OUTCOMES:
Best corrected visual acuity | 2 weeks after each laser session, 1, 2 and 3 months after pan-retinal photocoagulation is completed

CONTACTS AND LOCATIONS:
Overall Officials: Dulce O Rascon-Vargas, Fellow, Principal Investigator — Asociación Para Evitar la Ceguera en México I.A.P.; Guadalupe Cervantes-Coste, Study Chair — Asociación Para Evitar la Ceguera en México I.A.P.; Jans Fromow-Guerra, Study Director — Asociación Para Evitar la Ceguera en México I.A.P.
Locations (2):
- Mexico (2):
  - Asociación Para Evitar la Ceguera en México I.A.P., Mexico City
  - Asociacion para Evitar la Ceguera en Mexico I.A.P., Mexico City